CLINICAL TRIAL: NCT07089979
Title: A Randomized Study of the Glunovo Real-Time Continuous Glucose Monitoring (CGM) Effectiveness on Metabolic Control in Patients With Type 2 Diabetes (T2D)
Brief Title: Effectiveness of Glunovo Real-Time Continuous Glucose Monitoring in Adults With Type 2 Diabetes
Acronym: GCR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Milan (Other)
Responsible Party: Principal Investigator, Paolo Fiorina, MD, Professor, University of Milan
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 0023448/2024
Record Dates: First submitted 2025-04-09; First posted 2025-07-29 (Actual); Last update posted 2025-07-29 (Actual); Status verified 2025-07

CONDITIONS: Glucose Monitoring, Continuous
Keywords: Type 2 diabetes; Continous Glucose Monitoring; Glycemia
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- subjects who will use the device object of the interventional study (Experimental): Participants randomized to this arm used the Glunovo Real-Time Continuous Glucose Monitoring (RT-CGM) system for 6 months.
  Interventions: Device: Glunovo CGM device
- subjects who will use their glucometer (control group) (Placebo Comparator): Capillary glucose monitoring using fingerstick glucometer as per standard care.
  Interventions: Device: BG-meter

INTERVENTIONS:
Device: Glunovo CGM device — Group 1 (Subjects that will use Glunovo CGM device) will be compared to Group 2 (subject that will use their glucometer)
  Arms: subjects who will use the device object of the interventional study
Device: BG-meter — BG-meter
  Arms: subjects who will use their glucometer (control group)

SUMMARY:
The study aims to evaluate the effectiveness of the novel Real-Time Continuous Glucose Monitoring (RT-CGM) system "Glunovo" in improving glycemic control and patient-reported outcomes in individuals with poorly controlled Type 2 Diabetes (T2D).

DETAILED DESCRIPTION:
This is a prospective, open-label, randomized controlled trial involving 165 adult patients with T2D recruited at the Fatebenefratelli-Sacco Hospital in Milan. Participants were randomized in a 1:1 ratio to either the intervention group (RT-CGM with Glunovo) or the control group (standard Self-Monitoring of Blood Glucose [SMBG] using conventional glucometers).

The primary outcome is the change in Glycated Hemoglobin (HbA1c) levels after 6 months of follow-up. Secondary outcomes include Continuous Glucose Monitoring (CGM)-derived metrics-such as Glucose Management Indicator (GMI), Time in Range (TIR), Time Above Range (TAR), and Time Below Range (TBR)-as well as patient well-being, assessed using the WHO-5 Well-Being Index and a satisfaction scale.

The study is designed to assess whether the Glunovo RT-CGM system can support better metabolic control and improve patient experience compared to conventional SMBG methods.

ELIGIBILITY:
Inclusion Criteria:

Diagnosis of Type 2 Diabetes (T2D) Age above 18 years Glycated Hemoglobin (HbA1c) between 7.5% and 11% On basal-bolus insulin, basal-oral combination therapy, or non-insulin antidiabetic therapy

Exclusion Criteria:

Pregnancy HbA1c > 11% or < 7.5% Diagnosis of Type 1 Diabetes, Latent Autoimmune Diabetes in Adults (LADA), Maturity Onset Diabetes of the Young (MODY), or other forms of hyperglycemia

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 260 (Actual)
Dates: Start 2024-01-01 (Actual); Primary Completion 2024-07-01 (Actual); Study Completion 2024-07-15 (Actual)

PRIMARY OUTCOMES:
changes in HbA1c levels | 6 months
  The primary outcome of the study was to evaluate changes in HbA1c levels after 6 months of RT-CGM use compared to baseline in both the intervention and control groups

CONTACTS AND LOCATIONS:
Overall Officials: Prof. Paolo Fiorina, Principal Investigator — University of Milan
Locations (1):
- ASST Sacco Fatebenefratelli, Milan, Milan, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lazzaroni E, Cimino V, Gandolfi A, Tinari C, Bucciarelli L, Morpurgo P, Ben Nasr M, Fiorina RM, Pastore I, Baruffaldi L, Losurdo F, D'Addio F, Zuccotti GV, Montefusco L, Rossi A, Lunati ME, Fiorina P. A Randomized Study of the Glunovo Real-time CGM Effectiveness in Individuals With Poorly Controlled Type 2 Diabetes. J Endocr Soc. 2026 Jan 12;10(2):bvaf165. doi: 10.1210/jendso/bvaf165. eCollection 2026 Feb. PMID 41551204